CLINICAL TRIAL: NCT04010175
Title: Cognitive Training in Early to Moderate Stages Alzheimer's Disease Patients: Contribution of Digital Remote Training
Brief Title: Digital Cognitive Remote Training in Alzheimer's Disease (MA-EIAD)
Acronym: DCRT-AD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment stopped for thesis defense. It was not possible to extend the period of inclusion to achieve the patient objective
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0881
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Alzheimer Disease
Keywords: Cognitive training; Distance training; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator)
  Interventions: Behavioral: Control - Cognitive training in a practitioner's office one time per week
- Experimental group 1 (Experimental): Moderate frequency cognitive distance training
  Interventions: Behavioral: Experimental group 1 - Cognitive training in a practitioner's office one time per week and cognitive distance training one time per week
- Experimental group 2 (Experimental): High frequency cognitive distance training
  Interventions: Behavioral: Experimental group 2 - Cognitive training in a practitioner's office one time per week and cognitive distance training four times per week

INTERVENTIONS:
Behavioral: Control - Cognitive training in a practitioner's office one time per week — Participant will perform 1-hour cognitive computer based training one time per week in a practitioner's office during 4 months (16 weeks of training = 16 hours of training). This training will include 10 short tasks of increasing difficulty. Performance of these tasks involve cognitive functions such as: executive functions, reasoning, auditive, visual and visuo-spatial memory, speed of processing, short-term memory and working memory. Thus the training aims to exercise all these cognitive functions.
  Arms: Control group
Behavioral: Experimental group 1 - Cognitive training in a practitioner's office one time per week and cognitive distance training one time per week — Participant will perform 1-hour cognitive computer based training one time per week in a practitioner's office and one time per week cognitive distance training in her/his place of residence, during 4 months (16 weeks of training = 32 hours of training).
  Arms: Experimental group 1
Behavioral: Experimental group 2 - Cognitive training in a practitioner's office one time per week and cognitive distance training four times per week — Participant will perform 1-hour cognitive computer based training one time per week in a practitioner's office and four times per week cognitive distance training in her/his place of residence during 4 months (16 weeks of training = 80 hours of training).
  Arms: Experimental group 2

SUMMARY:
Cerebral functioning changes with age in order to respond to the impacts of different external and internal factors on the brain, and more generally on the human body. Scaffolding Theory of Aging and Cognition proposes that during life the brain develops specific neural networks to handle with cognitive activities. When these networks are impaired due to factors that damage brain structure and/or brain functioning, the brain adapts and elaborates new networks to cope with this situation. A cognitive reserve built throughout life and an appropriated care such as for example cognitive training, are in the centre of this model because they are involved in building these networks. In general, studies exploring cognitive training in normal aging and in patients suffering from neurodegenerative disease such as Alzheimer's disease have shown some benefits of the training on cognitive functioning. It has been shown not only that the cognitive training improves older adults' cognition, but also that these effects last for a long time and positively influence older people everyday activities. In fact, the benefits from memory training were observed 5 years after the end of the training and those of reasoning and of speed of processing even after 10 years. In addition, majority of the participants declared to notice improvement of their everyday life. Concerning Alzheimer's disease, several studies have observed positive results of cognitive training although there are some controversies about its' effects. Numerous studies point out that for cognitive training being the most efficient, the intervention has to take place as early as possible, preferentially in a premorbid stage of the disease and that it is important to propose trainings that minimize the withdrawal. In this sense, the importance of using computer based training was put forward because it allows the elaboration of multiple exercises with playful aspect and more importantly it can adapt on line the difficulty of the exercises to the patient's performance. However, if it is commonly admitted that computer based training has an important role in physician's, psychologist's or speech therapist's office less is known about the efficiency of this type of training performed at distance, at the patient's place of residence. It seems probable that to propose distance training as an additional training to that performed in a practitioner's office would increase training benefits. To investigators knowledge this was not investigated in a systematic way with Alzheimer's disease patients. The more important advantages of a such additional training are: (1) reduction of patients' travelling, (2) increased flexibility of training scheduling and (3) increased frequency of training sessions per week.

Thus, in the present study investigators will examine in a systematic way, whether the distance training, as an additional training to this performed in practitioner's office, brings incremental short- and long-term benefits coming from cognitive training in mild to moderate Alzheimer's disease patients. Investigators second objective is to determine what would be the best frequency per week of such an additional training.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more
* native French speaker
* Diagnosis of Alzheimer's disease according DMS-V criteria
* early to moderate stage of the disease (MMSE > 15)
* psychotropic drug treatment without change for three months at least
* signed informed consent
* being affiliated to a social security

Exclusion Criteria:

* not corrected visual or auditory deficit
* motor deficits preventing experimental tests execution
* ongoing participation in cognitive training or stimulation for more than three months
* not having a computer at the place of residence
* refusal of participation
* being under guardianship

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Influence of the training on experimental tasks | 8 months
  To evaluate benefits of cognitive training the scores of four experimental tasks will be combined.
  1. Stop Signal - inhibition score range 0 to 24, the higher values indicating better outcomes
  2. Updating Span - range 0 to 12, the higher values indicating better outcomes
  3. Letter-Number Pairs - flexibility score range 0 to 33, the higher values indicating better outcomes
  4. Operating Span - range 0 to 8, the higher values indicating better outcomes
Influence of the training on neuropsychological tests | 8 months
  To evaluate benefits of cognitive training the scores of five neuropsychological tests will be combined.
  1. Verbal Fluency - for letter P and animals, 0 to no limits; the higher values indicating better outcomes
  2. Trial Making Test A and B - reaction time in ms - the higher values indicating worse outcomes; number of errors - the higher values indicating better outcomes
  3. Logical Stories (MEM IV) - immediate memory score (0 to 53); - delayed memory score (0 to 50); - recognition score (0 to 30); the higher values indicating better outcomes.
  4. Mini mental State Examination (MMSE) - score from 0 to 30 (higher values indicating better outcomes)
  5. Verbal span (Wechsler Adult Intelligence Scale) - forward from 0 to 9 and backward from 0 to 8, the higher values indicating better outcomes
Influence of the training on global quality of life | 8 months
  To evaluate benefits of cognitive training scores of 6 questionnaires will be combined.
  1. Geriatric Depression Scale-0 to 30 (lower values indicating better outcomes)
  2. Questionnaire of Cognitive Complaint-0 to 10, higher values indicating worse outcomes
  3. Instrumental Activities of Daily Living-8 to 31, higher values indicating lower outcomes
  4. Pittsburgh Sleep Quality Index-0 (no difficulty) to 3(severe difficulty). Total score (summed)=0 to 21 (higher values indicating worse outcomes)
  5. SF-12 (questionnaire of quality of life)
  6. Motivational Scale for Older Adults-6 subscales of activities: Health; Related to biological needs ; Related to relationships with others; Related to religion; Related to leisure; Related to Information; For each subscales 4 motivation scores : 1) Extrinsic (0 to 21); 2) Amotivation (0 to 21); 3) Extrinsic - non self-detremined (0 to 21); 4) Intrinsic (0 to 21) The higher values indicating the higher level of each type of motivation/amotivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neuropsychologie - Hôpital Neurologique, Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimachki S, Tarpin-Bernard F, Croisile B, Chainay H. Study design and protocol of a low to high intensity computer-based cognitive training at home in supplement to standard care in patients with AD. BMJ Open. 2022 Jun 20;12(6):e050993. doi: 10.1136/bmjopen-2021-050993. PMID 35725247